CLINICAL TRIAL: NCT02018783
Title: Clinical Evaluation of the Effectiveness of Immediate Relief Obtained With Desensitizing Creams - A Controlled, Randomized, Triple Masked, Split-Mouth Clinical Trial
Brief Title: Single Application of Desensitizing Pastes as Dentin Sensitivity Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Olga Flecha, PhD, Federal University of São Paulo
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: dessensibilizantes
Record Dates: First submitted 2013-12-07; First posted 2013-12-23 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Dentine Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Sodium Fluoride; Sensodyne

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- Sensodyne (Experimental): Digital application for 60 seconds.
  Interventions: Procedure: Sensodyne
- Colgate (Experimental): Slow-speed handpiece with a Robson brush for 3 seconds by repeating the procedure
  Interventions: Procedure: Colgate
- Nano P (Experimental): Slow-speed handpiece with a Robson brush for 10 seconds
  Interventions: Procedure: Nano P
- Cocorico (Placebo Comparator): Digital application for 60 seconds
  Interventions: Procedure: Cocorico

INTERVENTIONS:
Procedure: Colgate — Slow-speed handpiece with a Robson brush for 3 seconds by repeating the procedure
  Arms: Colgate
Procedure: Sensodyne — Digital application for 60 seconds.
  Arms: Sensodyne
Procedure: Nano P — Slow-speed handpiece with a Robson brush for 10 seconds
  Arms: Nano P
Procedure: Cocorico — Digital application for 60 seconds
  Arms: Cocorico

SUMMARY:
The aim of this study was to evaluate the efficacy of three desensitizing toothpastes for immediate and intermediate-term relief of CDH, when compared with a control toothpaste. One hundred and thirty-eight hypersensitive teeth were diagnosed and randomized into four groups according to the therapeutic agent of each desensitizing cream tested: 1) strontium acetate and calcium carbonate, 2) calcium carbonate and arginine 8%, 3) calcium phosphate nanoparticles and 4) a control toothpaste. The desensitizing creams were applied according to the manufacturer's instructions. Cervical dentin hypersensitivity was assessed at baseline, immediately, 24 hours and 30 days after the treatment. Cold and evaporative tests were used to assess the sensitivity level.

ELIGIBILITY:
Inclusion Criteria:

* subjects 18 years or older
* in good general and oral health; have complaint of CDH in teeth distributed in all 4 quadrants
* not making use of desensitizing agents
* not having undergone periodontal treatment over the past 3 months
* respond to evaporative stimulus with a score ≥ 1.5 cm on VAS

Exclusion Criteria:

* patients who presented restorations and caries near the exposed dentin of the hypersensitive teeth
* who made frequent use of painkillers, anti-inflammatory and antidepressants drugs

Ages: 22 Years to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2013-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
cervical dentin hypersensitivity | 30 days
  The cervical dentin hypersensitivity was evaluated by an air blast (evaporative stimulus) for 5 seconds, and by a tetrafluoroethane spray (cold stimulus) for 5 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Olga D Flecha, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Periodontics Clinic, Department of Dentistry, Diamantina, Minas Gerais, Brazil